CLINICAL TRIAL: NCT06516003
Title: Use of Immersive Virtual Reality for Laceration Repairs in the Pediatric Emergency Department
Brief Title: VR for Lac Repairs in Peds Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29-01-FB-0211
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Laceration
Keywords: virtual reality; pediatrics; emergency department
MeSH Terms: conditions — Lacerations; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Patients randomized to receive virtual reality goggles in addition to the standard of care.
  Interventions: Device: Immersive Virtual Reality Goggles
- Standard of Care (Active Comparator): Patients that are randomized to receive the standard of care including other distraction techniques and child life specialist.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Device: Immersive Virtual Reality Goggles — Immersive Virtual Reality goggles are a head mounted device placed over a patient's head and eyes that allows them to play in a virtual reality game.
  Arms: Virtual Reality
Behavioral: Standard of Care — Distraction techniques like tablet, phone, television, parent, child life specialist
  Arms: Standard of Care

SUMMARY:
The goal of the clinical trial is to compare virtual reality to standard of care for laceration repairs in the pediatric emergency department. The main question it aims to answer is:

-Does virtual reality decrease pain and anxiety scores compared to standard of care for laceration repairs in the pediatric emergency department?

Participants who meet the age and other inclusion criteria will be enrolled by research staff. They will complete a brief paper survey along with their guardians and the provider doing the laceration repair. The surveys will be completed after the laceration repair is finished.

DETAILED DESCRIPTION:
This will be a randomized pragmatic study for all patients ages 6-17 years with simple lacerations. Simple lacerations will be defined as lacerations within the scope of pediatric emergency medicine providers AND not requiring sedation or operative intervention. Subjects will be identified by the Emergency Department staff for enrollment. The goal number of enrolled participants will be 480, including 240 patients randomized into two groups, 120 per group, and 240 parents/guardians. The Emergency Department accepted to participate in this study and ED providers will complete the provider's survey. After signing the consent and assent form when appropriate, the patients will be randomized to either receive the standard of care or standard or care with immersive virtual reality goggles. Consent and assent will be obtained in the patient rooms within the emergency department. The standard of care shall be defined to include any of the following: local analgesia (topical LET and/ or subcutaneous lidocaine), oral or intranasal midazolam, distraction, Child Life Staff, or physical holding. Because each of the aforementioned interventions may vary between patients, it cannot be truly standardized; hence, this will be considered a pragmatic study. Patients randomized to the VR arm will receive the other standard procedures as well with VR goggles as an adjunct. Exclusion criteria include a history of epilepsy, visual or hearing impairment, or intellectual disability that would preclude use of VR goggles as determined by the guardian. Additionally, any lacerations around the eyes, eyebrows, and nose will be excluded as well as patients requiring sedation. Non-English speaking patients will be excluded as well. Hand lacerations will not be excluded.

Participants will be identified by ED staff following evaluation of the laceration. The ED staff will be given a flowchart with eligibility criteria. All interested participants who meet eligibility criteria will be consented. A research team member will obtain consent from parents or guardians by providing and reviewing the consent form (see Subject Consent Form). For patients who are between 8 and 17 years of age, a research team member will obtain assent by providing and reviewing the assent form (see Subject Assent Form). Consent and assent will be obtained in the patient's ED room.

Patients will be separated into groups age 6-11 and 12-17. Patients will be randomized via a selection of a sealed envelope which will contain instructions for use of the VR goggles. The goggles utilized will be Lenovo Mirage Solo with DayDream, which are standalone VR headset with Worldsense Body Tracking. Research staff will coach the child on age-appropriate games, as previously determined by Lenovo.

The goggles will be cleansed with Oxivir Tb disinfectant wipes after each use and allowed to dry in room air prior to next use. Education will be provided to all ED providers on the proper cleansing protocol for the VR goggles (Figure 4). The disinfectant protocol will be available for all users during the study, and has been approved by the director of Infection Control at Children's Hospital of the King's Daughters.

Following the laceration repair, the patient, guardian and health care provider will be surveyed (Figure 1, 2, and 3) on paper surveys. The survey includes Likert-type scale questions, binary questions as well as incorporates the Wong Baker Faces Pain Scale and Children's Fear Scale. The duration of the procedure will be recorded by the healthcare provider who completed the laceration repair. Time of procedure will be defined as from the time of irrigation to wound dressing. Patients and parents will both be filling out their own individual surveys. The parent should complete the survey first before the child should the child need assistance with completion. Patients and parents may decline to participate in any survey at any time

ELIGIBILITY:
Inclusion Criteria:

* Simple lacerations that do not require surgical subspecialty repair or moderate or deep sedation
* Hand lacerations
* Laceration that required stitches

Exclusion Criteria:

* less than 6 years old or greater than 17 years old
* Non english speaking
* Visual or hearing impairment
* Epilepsy
* Lacerations to forehead, nose, or cheeks where goggles cover
* Intellectual disability that precludes participation as determined by guardian

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Pain Score | Assessed immediately after intervention
  Using Wong Baker Faces Pain Scale
Fear Score | Assessed immediately after intervention
  Using Children's Fear Score

SECONDARY OUTCOMES:
Satisfaction of procedure | Assessed immediately after intervention
  Assessed by Likert- type scale question
Side Effects | Assessed immediately after intervention
  nausea, vomiting, dizziness, headache, other
Duration of procedure | Assessed immediately after intervention
  Five minute intervals up to 25 minutes
Future Use | Assessed immediately after intervention
  Would they recommend use of VR for same procedure again
Physical Holding | Assessed immediately after intervention
  Did patient need to be held for the procedure
Anxiolytic Use | Assessed immediately after intervention
  Did patient need anxiolytics for the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Not planning to share data with other researchers

REFERENCES:
- [Background] Martin SR, Heyming TW, Fortier MA, Kain ZN. Paediatric laceration repair in the emergency department: post-discharge pain and maladaptive behavioural changes. Emerg Med J. 2024 Jul 22;41(8):469-474. doi: 10.1136/emermed-2023-213858. PMID 38724104
- [Background] Ploghaus A, Narain C, Beckmann CF, Clare S, Bantick S, Wise R, Matthews PM, Rawlins JN, Tracey I. Exacerbation of pain by anxiety is associated with activity in a hippocampal network. J Neurosci. 2001 Dec 15;21(24):9896-903. doi: 10.1523/JNEUROSCI.21-24-09896.2001. PMID 11739597
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Kumar K, Ali S, Sabhaney V, Trottier E, Drendel A, Bhatt M, Boisvert L, Poonai N; Pediatric Emergency Research Canada. Anxiolysis for laceration repair in children: a survey of pediatric emergency providers in Canada. CJEM. 2022 Jan;24(1):75-83. doi: 10.1007/s43678-021-00210-y. Epub 2021 Nov 8. PMID 34746980
- [Background] Ali S, McGrath T, Drendel AL. An Evidence-Based Approach to Minimizing Acute Procedural Pain in the Emergency Department and Beyond. Pediatr Emerg Care. 2016 Jan;32(1):36-42; quiz 43-4. doi: 10.1097/PEC.0000000000000669. PMID 26720064
- [Background] Arikan A, Esenay FI. Active and Passive Distraction Interventions in a Pediatric Emergency Department to Reduce the Pain and Anxiety During Venous Blood Sampling: A Randomized Clinical Trial. J Emerg Nurs. 2020 Nov;46(6):779-790. doi: 10.1016/j.jen.2020.05.004. Epub 2020 Jul 22. PMID 32711948
- [Background] Aykanat Girgin B, Gol I. Reducing Pain and Fear in Children During Venipuncture: A Randomized Controlled Study. Pain Manag Nurs. 2020 Jun;21(3):276-282. doi: 10.1016/j.pmn.2019.07.006. Epub 2019 Sep 26. PMID 31501078
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] Arane K, Behboudi A, Goldman RD. Virtual reality for pain and anxiety management in children. Can Fam Physician. 2017 Dec;63(12):932-934. PMID 29237632
- [Background] Piskorz J, Czub M. Effectiveness of a virtual reality intervention to minimize pediatric stress and pain intensity during venipuncture. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12201. Epub 2017 Nov 20. PMID 29155488
- [Background] Thomas JJ, Albietz J, Polaner D. Virtual reality for lumbar puncture in a morbidly obese patient with leukemia. Paediatr Anaesth. 2018 Nov;28(11):1059-1060. doi: 10.1111/pan.13505. Epub 2018 Oct 4. PMID 30284748
- [Background] Hoffman HG, Rodriguez RA, Gonzalez M, Bernardy M, Pena R, Beck W, Patterson DR, Meyer WJ 3rd. Immersive Virtual Reality as an Adjunctive Non-opioid Analgesic for Pre-dominantly Latin American Children With Large Severe Burn Wounds During Burn Wound Cleaning in the Intensive Care Unit: A Pilot Study. Front Hum Neurosci. 2019 Aug 8;13:262. doi: 10.3389/fnhum.2019.00262. eCollection 2019. PMID 31440148
- [Background] Chad R, Emaan S, Jillian O. Effect of virtual reality headset for pediatric fear and pain distraction during immunization. Pain Manag. 2018 May;8(3):175-179. doi: 10.2217/pmt-2017-0040. Epub 2018 May 3. PMID 29722606
- [Background] Shetty V, Suresh LR, Hegde AM. Effect of Virtual Reality Distraction on Pain and Anxiety During Dental Treatment in 5 to 8 Year Old Children. J Clin Pediatr Dent. 2019;43(2):97-102. doi: 10.17796/1053-4625-43.2.5. Epub 2019 Feb 7. PMID 30730798
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326
- [Background] Goldman RD, Behboudi A. Pilot Randomized Controlled Trial of Virtual Reality vs. Standard-of-Care During Pediatric Laceration Repair. J Child Adolesc Trauma. 2021 Mar 26;14(2):295-298. doi: 10.1007/s40653-021-00350-4. eCollection 2021 Jun. PMID 33986914
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Bexson C, Oldham G, Wray J. Safety of virtual reality use in children: a systematic review. Eur J Pediatr. 2024 May;183(5):2071-2090. doi: 10.1007/s00431-024-05488-5. Epub 2024 Mar 11. PMID 38466416
- [Background] Neiman NR, Falkson SR, Rodriguez ST, Wang EY, Hemphill SF, Khoury ME, Kist MN, Jackson CD, Caruso TJ. Quantifying virtual reality pain modulation in healthy volunteers: A randomized, crossover study. J Clin Anesth. 2022 Sep;80:110876. doi: 10.1016/j.jclinane.2022.110876. Epub 2022 May 4. PMID 35525050
- [Derived] McEvoy AO, Vincent OB, Vazifedan T, Chang TP, Clingenpeel JM, Kapoor R. Virtual Reality as Active Distraction in Laceration Repair: A Game Changer? Pediatr Emerg Care. 2025 Mar 1;41(3):208-212. doi: 10.1097/PEC.0000000000003319. Epub 2024 Dec 6. PMID 39641640

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT06516003/Prot_SAP_000.pdf